CLINICAL TRIAL: NCT06653790
Title: EFFECT of PSYCHOSOCIAL STIMULATIONS on TREATMENT OUTCOME of SEVERE ACUTE MALNOURISHED CHILDREN
Brief Title: PSYCHOSOCIAL STIMULATIONS and TREATMENT OUTCOME of SEVERE ACUTE MALNOURISHED CHILDREN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BMU-HS
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Malnutrition Severe

STUDY DESIGN:
Intervention Model Description: The severely acute malnourished children in intervention group will be sent to development pediatrician who will do a developmental assessment of the child and stimulation. A sensory therapist, an occupational and a physiotherapist will also be available for sessions. The psychosocial stimulation will be offered in two phases: in-patient (at stabilization unit) and after discharge, patient will be referred to outpatient (at outpatient therapeutic center) and developmental outpatient. The sessions with development pediatrician and team will be held every week lasting for about 20-40 min in the presence of the caregiver. The intervention includes auditory, tactile and visual stimulation, hand-eye coordination, and different types of sensory-motor training that include fine and gross motor activities. The guiding principle will be to enhance a child's holistic development-cognitive, language, physical, and social-in an integrated manner by using age-appropriate play materials, cultural t
Who Masked: Care Provider, Investigator
Masking Description: The care provider and investigators will be blided
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): The psychosocial stimulation will be offered in two phases: in-patient (at stabilization unit) and after discharge patient will be referred to out-patient (at outpatient therapeutic centre) and developmental out-patient. The sessions with development paediatrician and team will be held every week lasting for about 20-40 min in the presence of the caregiver. The intervention includes auditory, tactile and visual stimulation, hand-eye coordination, and different types of sensory-motor training that included fine and gross motor activities. The guiding principle will be to enhance a child's holistic development-cognitive, language, physical, and social-in an integrated manner by using age-appropriate play materials, cultural tools, and resources.
  Interventions: Behavioral: Psychosocial stimulations
- Control (No Intervention): The control arm will be given no intervention except standard treatment

INTERVENTIONS:
Behavioral: Psychosocial stimulations — The psychosocial stimulation will be offered in two phases: in-patient (at stabilization unit) and after discharge patient will be referred to out-patient (at outpatient therapeutic centre) and developmental out-patient. The sessions with development paediatrician and team will be held every week lasting for about 20-40 min in the presence of the caregiver. The intervention includes auditory, tactile and visual stimulation, hand-eye coordination, and different types of sensory-motor training that included fine and gross motor activities. The guiding principle will be to enhance a child's holistic development-cognitive, language, physical, and social-in an integrated manner by using age-appropriate play materials, cultural tools, and resources.
  Arms: Intervention arm

SUMMARY:
A playroom and a playground are already part of the stabilization unit and are furnished with basic facilities for engaging the SAM children in play-based motor, language, and personal-social activities. The severely acute malnourished children in the intervention group will be sent to a development pediatrician who will do a developmental assessment of the child and stimulation. A sensory therapist, an occupational therapist, and a physiotherapist will also be available for sessions.

DETAILED DESCRIPTION:
The World Health Organisation (WHO) also suggests including psychological stimulation in the treatment of severe acute malnutrition. However, there is limited evidence that these interventions are beneficial for SAM children, especially when there are severe food shortages and a lack of a balanced diet.

There is limited available research in Pakistan examining the impact of psychosocial stimulation on severely malnourished children and a significant gap in its implementation. It is obvious that current implementation research is needed to understand how to improve brain development in children with SAM who require inpatient care in a practical and pragmatic approach.

The purpose of this study is to present data on the efficacy of these therapies, which may help shape future SAM treatment plans and policies. Mitigating the physical and mental dimensions of malnourishment can result in more enduring and significant consequences, ultimately enhancing the standard of living for millions of children around the globe.

ELIGIBILITY:
Inclusion Criteria:

* All children aged 6m to 59 months admitted to stabilization centre fulfilling criteria of severe acute malnutrition will be included in study.

Exclusion Criteria:

* Children with chronic diseases like cystic fibrosis, cerebral palsy, celiac disease, chronic kidney disease, chronic liver failure, congenital heart disease, inborn error of metabolism, cleft lip and palate will be excluded from study.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Developmental performance | 6- months from baseline
  Developmental performance in terms of gross motor, fine motor, language and personal-social by using Denver II developmental screening test. The number of test items that a child has successfully performed (passed) is described as the performance score. A child is delayed if he fails to perform what 90% of children of that age can perform. Caution is raised if a child is not able to perform a task that 75% to 90% of children can perform.

SECONDARY OUTCOMES:
Child growth | 6- months from baseline
  Growth in terms of z-scores (improved from < -- 3 to < --1 z-score) and MUAC ( improved from < 11.5 cm to > 12.5 cm).

IPD SHARING:
Plan to Share IPD: No
Methodology, statistical plan, and results will be published in peer-reviewed journals

REFERENCES:
- [Background] Nahar B, Hamadani JD, Ahmed T, Tofail F, Rahman A, Huda SN, Grantham-McGregor SM. Effects of psychosocial stimulation on growth and development of severely malnourished children in a nutrition unit in Bangladesh. Eur J Clin Nutr. 2009 Jun;63(6):725-31. doi: 10.1038/ejcn.2008.44. Epub 2008 Sep 3. PMID 18772893
- [Background] Yousafzai AK, Obradovic J, Rasheed MA, Rizvi A, Portilla XA, Tirado-Strayer N, Siyal S, Memon U. Effects of responsive stimulation and nutrition interventions on children's development and growth at age 4 years in a disadvantaged population in Pakistan: a longitudinal follow-up of a cluster-randomised factorial effectiveness trial. Lancet Glob Health. 2016 Aug;4(8):e548-58. doi: 10.1016/S2214-109X(16)30100-0. Epub 2016 Jun 21. PMID 27342433
- [Background] Worku BN, Abessa TG, Wondafrash M, Vanvuchelen M, Bruckers L, Kolsteren P, Granitzer M. The relationship of undernutrition/psychosocial factors and developmental outcomes of children in extreme poverty in Ethiopia. BMC Pediatr. 2018 Feb 9;18(1):45. doi: 10.1186/s12887-018-1009-y. PMID 29426302
- [Background] Ethiopian FMoH. Job aid for maternal nutrition and age Appropriate Infant & Young Child Nutrition: Addis Ababa; 2016.